CLINICAL TRIAL: NCT00738322
Title: A Single-Centre, Single-Blind, Randomised, Placebo-Controlled, Phase I Study to Assess the Safety, Tolerability and Pharmacokinetics After Single Ascending Intravenous Doses of AZD1305 in Healthy Male Japanese Subjects
Brief Title: To Study Safety, Tolerability and Pharmacokinetics of AZD1305 in Healthy Male Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Helen Lunde, MD, Medical Science Director, Emerging Arrhythmias & Lipids, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D3191C00001
Record Dates: First submitted 2008-07-11; First posted 2008-08-20 (Estimated); Last update posted 2009-06-30 (Estimated); Status verified 2009-06

CONDITIONS: Healthy
Keywords: AZD1305; safety; pharmacokinetics; single ascending doses; Japanese; male
MeSH Terms: interventions — tert-butyl (2-(7-(2-(4-cyano-2-fluorophenoxy)ethyl)-9-oxa-3,7-diazabicyclo(3.3.1)non3-yl)ethyl)carbamate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: AZD1305
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD1305 — Solution for iv infusion, single dose
  Arms: 1
Drug: Placebo — NaCl solution for iv infusion, single dose
  Arms: 2

SUMMARY:
The purpose is to study the safety of AZD1305, how AZD1305 is tolerated and how the medication is metabolised by the body ( how it is taken up into the body, distributed around the body and disappears from the body) in healthy Japanese males.

ELIGIBILITY:
Inclusion Criteria:

* A body mass index (BMI=weight/height2) of 19 to 27 kg/m2
* Japanese males

Exclusion Criteria:

* ECG findings outside normal reference ranges.
* Potassium outside normal reference ranges.

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2008-07; Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Safety by assessment of adverse events, ECG variables, BP, pulse rate, physical examination, laboratory variables, body temperature and body weight | During the study

SECONDARY OUTCOMES:
Pharmacokinetic variables | During the dosing visits

CONTACTS AND LOCATIONS:
Overall Officials: Helen Lunde, MD, Study Director — AstraZeneca R&D, Mölndal, Sweden; Kyoko Matsuguma, MD, Principal Investigator — Kyushu Clinical Pharmacology Research Clinic, Fukuoka, Japan
Locations (1):
- Research Site, Fukuoka, Japan